CLINICAL TRIAL: NCT02165644
Title: Targeting Carbonic Anhydrase Mediated Coupling as a Novel Vasospasm Prophylaxis in Aneurysmal Sub Arachnoid Hemorrhage
Brief Title: Carbonic Anhydrase Antagonism in Subarachnoid Hemorrhage
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The PI is leaving the University of Florida.
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014000419
Record Dates: First submitted 2014-06-13; First posted 2014-06-17 (Estimated); Last update posted 2015-09-24 (Estimated); Status verified 2015-09

CONDITIONS: Acute Cerebrovascular Accident; Vasospasm
Keywords: Subarachnoid Hemorrhage; Vasospasm; Acetazolamide
MeSH Terms: conditions — Stroke; Subarachnoid Hemorrhage | interventions — Acetazolamide; Nimodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Acetazolamide (Experimental): Acetazolamide 250 mg QID oral for 4 days along with current standard of care which is Nimodipine 60 mg orally every 4 hours, with therapy starting within 96 hours of the event and continued for 21 days.
  If the drug can't be given orally, then feeding tube (NG Tube or DHT) will be used for drug administration.
  Interventions: Drug: Acetazolamide; Drug: Nimodipine
- Standard of care (Active Comparator): Subjects will receive only standard of care for subarachnoid hemorrhage which will include Nimodipine 60 mg orally every 4 hours, with therapy starting within 96 hours of the event and continued for 21 days.
  Interventions: Drug: Nimodipine

INTERVENTIONS:
Drug: Acetazolamide — Acetazolamide 250 mg QID oral for 4 days along with standard of care which includes Nimodipine 60 mg orally every 4 hours, with therapy starting within 96 hours of the event and continued for 21 days.
  If the drug can't be given orally, then feeding tube (NG Tube or DHT) will be used for drug administration.
  Other Names: Diamox
  Arms: Acetazolamide
Drug: Nimodipine — Nimodipine 60 mg orally every 4 hours, with therapy starting within 96 hours of the event and continued for 21 days
  Other Names: Nimotop

SUMMARY:
Subarachnoid Hemorrhage (SAH) can occur commonly in the setting of trauma or brain aneurysm. SAH accounts for 10% of all the strokes. Aneurysmal SAH accounts for 80 % of cases of non-traumatic cases of SAH, 6-8% of all strokes and 22-25% of all cerebrovascular deaths. Mortality can be 50% in the first few years of aneurysmal SAH rupture, 15% are severely disabled post SAH and only 20-35% having a moderate to good recovery it has gained lot of attention and pre-clinical and clinical trials of various agents have been tried to prevent poor outcome. The United States epidemiology data reveals the fact that 1% to 5% of adults have unruptured brain aneurysm and 30,000 people suffer from aneurysm rupture annually translating to brain aneurysm rupture every 18 minutes.

Vasospasm is the most common SAH complication post 24 hours. It is the segmental or diffuse narrowing of the vessels especially the large vessels. Fifty percent of those patients who develop clinical vasospasm, progress to infarction and 15-20% will advance to disabling stroke or die of cerebral ischemia. The present treatment modalities are insufficient to prevent vasospasm. So, we need new treatment modalities to decrease the mortality and morbidity in SAH patients.

The investigators hypothesize that Acetazolamide administration can prevent development of vasospasm after aneurysmal SAH.

DETAILED DESCRIPTION:
If the subject decides to take part in this study, they will receive acetazolamide with standard of care or standard of care only for four days. This means:

The subject will be given acetazolamide tablet orally with standard care for subarachnoid hemorrhage or standard of care only, for a maximum of 4 days. If the subject cannot take medication orally then the investigators will put a tube through the nose to stomach or small intestine. Being part of the study does not exclude the subject from receiving the standard therapy. The subject will be given the current standard of care therapy irrespective of being in the study or not. The investigators will review the subject's medical records and collect information from standard of care procedures that would have been done even if the subject were not enrolled in this study. This information will include, but will not be limited to, the subject's imaging data, sub arachnoid hemorrhage assessments and medical history. The subject's Hunt and Hess scale score and (World federation of neurologic surgeons) WFNS scale score will also be collected. Hunt and Hess and WFNS scale are used to assess the level of damage to neurologic functions of a person caused by sub arachnoid hemorrhage.

The subject will be asked to come for the follow-up at 3 months after the discharge from the hospital. The following data will be obtained from each subject at 3-month follow-up.

1. Modified Rankin Scale (m-RS) scores
2. Glasgow Outcome Scale (GOS) scores

ELIGIBILITY:
Inclusion Criteria:

1. All aneurysmal SAH patients with clinical and or radiological diagnosis.
2. Subjects with age ≥18 years and ≤80 years at the time of screening.
3. The subject or his/ her legal representative is willing to undergo informed consent process prior to enrollment into this study.
4. World Federation of Neurosurgeons scale score ≤ 2
5. Hunt and Hess Stroke scale score ≤ 2
6. Mean velocities of < 200 cm/s in at least 1 vascular axis of the circle of Willis
7. Patients admitted within 4 days of symptom onset.

Exclusion Criteria:

1. Subject with age < 18 years and >80 years at the time of screening.
2. Time of symptom onset cannot be determined.
3. Subject who is pregnant or lactating.
4. Subjects who have hypersensitivity to acetazolamide, sulfa drugs, or any component of the formulation.
5. Mean velocities of ≥ 200 cm/s in at least 1 vascular axis of the circle of Willis
6. Brain CT or MRI show acute infarction
7. Any acute focal neurological deficit (including any one of these) speech problems, loss of vision, facial or extremity weakness.
8. Hunt and Hess Stroke scale scores > 2
9. World Federation of Neurosurgeons scale scores > 2
10. Subjects with hepatic disease or insufficiency or cirrhosis.
11. Subjects with severe renal disease or dysfunction.
12. Subjects who have decreased sodium and/or potassium levels; hyperchloremic acidosis.
13. Subjects who have adrenocortical insufficiency.
14. The subject or legal representative is unable to provide informed consent.
15. The subject is medically unstable to participate in the trial as determined by the principal investigator.
16. The subject has any end stage medical condition as determined by the principal investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Score | At 3 months from the baseline
  The modified Rankin Scale (m-RS) is a commonly used scale for measuring the degree of disability or dependence in the daily activities of people after they have suffered a stroke including subarachnoid hemorrhage. The score is given according to following scale.
  0- No symptoms at all
  1. No significant disability despite symptoms; able to carry out all usual duties and activities
  2. Slight disability; unable to carry out all previous activities, but able to look after own affairs without assistance
  3. Moderate disability; requiring some help, but able to walk without assistance
  4. Moderately severe disability; unable to walk without assistance and unable to attend to own bodily needs without assistance
  5. Severe disability; bedridden, incontinent and requiring constant nursing care and attention
  6. Dead
Neurological examination of the subject | Baseline, 10 days, 3 months
  Neurological status of a subject is assessed by physical neurological examination of the subject by a qualified neurologist. It is one of the most important aspect in determining neurological health of a subject after subarachnoid hemorrhage. It also helps to determine subarachnoid hemorrhage severity and prognosis.
Glasgow Outcome Score | At 3 months from the baseline
  The Glasgow Outcome Scale (GOS) was developed to rank outcomes after head injury, but has been used in stroke studies including subarachnoid hemorrhage. The score is given according to following scale ranging from 1-5.
  1. Death- Severe injury or death without recovery of consciousness
  2. Persistent vegetative state- Severe damage with prolonged state of unresponsiveness and a lack of higher mental functions
  3. Severe disability- Severe injury with permanent need for help with daily living
  4. Moderate disability- No need for assistance in everyday life, employment is possible but may require special equipment.
  5. Low disability- Light damage with minor neurological and psychological deficits.
Hunt and Hess Scale | Baseline, 10 days
  The Hunt and Hess scale, is one of the grading systems used to classify the severity of a subarachnoid hemorrhage based on the patient's clinical condition. It is used as a predictor of patient's prognosis/outcome, with a higher grade correlating to lower survival rate. It gives an index of the mortality associated with the various grades. The mortality is minimum with grade 1 and maximum with grade 5. The grades are as follows:
  1. Asymptomatic, mild headache, slight nuchal rigidity
  2. Moderate to severe headache, nuchal rigidity, no neurologic deficit other than cranial nerve palsy
  3. Drowsiness / confusion, mild focal neurologic deficit
  4. Stupor, moderate-severe hemiparesis
  5. Coma, decerebrate posturing
World Federation of Neurosurgeons Scale | Baseline, 10 days
  The World Federation of Neurosurgeons (WFNS) classification uses Glasgow coma score (GCS) and focal neurological deficit to gauge severity of symptoms. It is intended to be a simple, reliable and clinically valid way to grade a patient with subarachnoid hemorrhage. The prognosis becomes worse when we move from grade 1 to grade 5.
  Grade 1 represents a GCS of 15 with absent focal neurological deficit, Grade 2 represents a GCS of 13-14 with absent focal neurological deficit, Grade 3 represents a GCS of 13-14 with focal neurological deficit present, Grade 4 represents a GCS of 7-12 with present or absent focal neurological deficit, Grade 5 represents a GCS of <7 with present or absent focal neurological deficit.

CONTACTS AND LOCATIONS:
Overall Officials: Vishnumurthy S Hedna, MD, Principal Investigator — University of Florida